CLINICAL TRIAL: NCT04811898
Title: A Dose Escalation Phase I Study of LNA-i-miR-221 for the Treatment of Refractory Multiple Myeloma and Advanced Solid Tumors
Brief Title: A Dose Escalation Study of LNA-i-Mir-221 for Cancer Treatment
Acronym: LNA-i-miR221
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Mater Domini, Catanzaro (Other)
Collaborators: Associazione Italiana per la Ricerca sul Cancro (Other)
Responsible Party: Principal Investigator, TASSONE PIERFRANCESCO, Professor of Medical Oncology, Magna Graecia University, Catanzaro, Italy, Azienda Ospedaliera Universitaria Mater Domini, Catanzaro
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AOU-MD FIH-LNA-i-miR-221; 2017-002615-33 (EudraCT Number)
Record Dates: First submitted 2021-02-27; First posted 2021-03-23 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Multiple Myeloma, Refractory; Hepatocarcinoma; Advanced Solid Tumor
Keywords: LNA-i-miR-221; Multiple Myeloma; Hepatocarcinoma; Advanced solid tumors; Phase I; Dose escalation; Safety; maximum tolerated dose (MTD); RP2D
MeSH Terms: conditions — Multiple Myeloma; Carcinoma, Hepatocellular | interventions — LNA-i-miR-221

STUDY DESIGN:
Intervention Model Description: monocentric, open label, phase I dose-escalation to determine the safety, the maximum tolerated dose (MTD) and the recommended phase II dose of LNA-i-miR-221 (RP2D) in a minimum/maximum number of 15/36 subjects affected by MM and advanced solid tumors. LNA-i-miR-221 will be administered IV daily infusion on days 1-4 followed by 24 days washout (1 cycle lasting 28 days) with a modified 3+3 Fibonacci dose escalation design, with 5 different dose levels for each cohort (0,5 mg/kg; 1 mg/kg; 2 mg/kg; 3 mg/kg; 5 mg/kg).
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental single arm (Experimental): Single group with 5 dose escalation for each cohort (0,5 mg/kg; 1 mg/kg; 2 mg/kg; 3 mg/kg; 5 mg/kg)
  Interventions: Biological: LNA-i-miR-221

INTERVENTIONS:
Biological: LNA-i-miR-221 — LNA-i-miR-221, IV daily infusion on days 1-4 followed by 24 days washout (1 cycle lasting 28 days)

SUMMARY:
The LNA-i-miR-221 Phase I trial has been designed as a monocentric open label dose escalation study which received written approval by the Competent Authority and independent Ethics Committee (IEC). LNA-i-miR-221 will be investigated for safety and tolerability in patients, men and women age ≥18 yrs, affected by Refractory-MM and advanced solid tumors.

DETAILED DESCRIPTION:
The LNA-i-miR-221 Phase I trial is a no-profit fully academic study on research funds and no external sponsor does exist. The study is a monocentric, open-label, phase I dose-finding to determine the safety, the maximum tolerated dose (MTD), and the recommended phase II dose of LNA-i-miR-221 (RP2D) using escalating doses; The secondary endopoints will be plasma and urinary pharmacokinetc (PK), efficacy as preliminary exploration of the antitumor activity, the disease control and the evaluation of biomonitoring activity. The study will include refractory MM and advanced solid tumors. In the last cohort, if 3 out of 3 or 5 out of 6 subjects do not experience DLT, no further dose escalation will be required and dose level 5 will be declared the MTD. At the end, further expansion will be performed to define RP2D, after a critical evaluation of trial data by SRC. LNA-i-miR-221 is a 13-mer antisense miR-221 inhibitor, which takes advantage of locked nucleic acid (LNA) technology and phosphorotioate (PS) backbone chemistry to increase affinity for miR-221 and nuclease resistance and represents a new frontier for chemically modified antisense oligonucleotides.

Participants will be assigned to 5 different cohorts, according to 5 different dose levels used. The cohorts will be defined with progressive numbers (1, 2, 3, 4, 5). Each cohort will be composed of 3 to 6 subjects. The dose level of LNA-i-miR-221 will be increased from one cohort to the next one. Independently from the assigned dose level, patients from each cohort will receive a total of 4 IV administrations as boluses. The treatment cycle will last 28 days. Each subject who will not experience any DLT (see DLT definition) will remain on the assigned dose level. In the case that MTD will be defined by the occurrence of DLT at the superior level, the MTD cohort will be considered for expansion to definitely assess the RP2D studies.

The treatment schedule (as amended and approved by AIFA on 1/15/2020) will be IV daily infusion on days 1-4 followed by 24 days washout (1 cycle lasting 28 days) with a modified 3+3 Fibonacci dose escalation design, with 5 different dose levels for each cohort (0,5 mg/kg; 1 mg/kg; 2 mg/kg; 3 mg/kg; 5 mg/kg), for safety and toxicity evaluation, MTD assessment, PK and modulatory activity investigation in refractory MM and advanced solid cancer patients. No other investigational drug and/or standard antitumor chemotherapy will be allowed during the study.

The enrolled subject will require hospitalization to ensure adequate protocol adherence.

LNA-i-miR-221will be administered inpatient setting as intravenous infusion of 30 minutes. During infusion and the following two hours post infusion, patients will be continuously monitored for vital signs. Local healthy authority guidelines must be followed with regard to further observation and monitoring, if applicable. Following the first infusion, patients will be observed for at least 120 minutes for fever, chills, or other infusion-associated symptoms. If prior infusions were well tolerated (without any signs or symptoms of infusion reactions) subsequent doses of LNA-i-miR-221 will be administered in 30 minutes with a 120 minutes observation period after infusion.

The determination of LNA-i-miR-221 in human plasma and urine will be used for the pharmacokinetic evaluation. For each enrolled subject, 2-5 ml of blood samples will be drawn for the quantification of LNA-i-miR-221 before, after 15 min and at the end of infusion at the following time points: 0.5, 1, 2, 4, 6, 12 hours on days 1 and 2. On day 3 and 4, blood samples will be drawn before and at the end of infusion at the following time points: 1, 2, 4. At 24 hours (day 5) and 48 hours (day 6) after last administration blood samples will be drawn for the quantification of LNA-i-miR-221.

Urine pharmacokinetic samples (15-20 ml) will be collected at pre-dose and 6, 12 and 24 hours period postdose on day 1 of cycle of treatment. Aliquots (15-20 ml) of 24-hour urine will also be collected at post dosing time during the cycle of treatment (day 2, 3, 4 and 5).

The vials containing lyophilized LNA-i-miR-221 must be stored at +2-8°C, while the reconstituted solution must be manipulated rapidly in a safe and secure place below 25°C, with no access for unauthorized personnel. The solution can be reconstituted immediately before administration. All adverse events will be followed with appropriate medical management until resolved. Patients removed from study for unacceptable adverse events will be followed until resolution or stabilization of the adverse event. For selected adverse events for which administration of the investigational drug was stopped, a rechallenge of the subject with the investigational drug may be conducted if considered both safe and ethical by the study coordinator.

All the safety data will be reviewed by an independent Safety Review Committee (SRC). Dose escalation to the next dose level will be allowed by SRC. In the last cohort, if 3 out of 3 or 5 out of 6 subjects do not experience DLT, no further dose escalation will be required and dose level 5 will be declared the MTD. At the end, further expansion will be performed to define RP2D, after a critical evaluation of trial data by SRC. At 30 (+/-1) days from the first dose of treatment, each enrolled patients will be evaluated for the end of treatment (EOT) visit in order to evaluate the efficacy and clinical benefit of LNA-i-miR-221 treatment based on RECIST V1.1 criteria. Only for patients with clinical benefit or radiological response/stable disease, the treatment will be offered until disease progression or if the patient withdraws consent. Out patients follow up will be continued every two months, until death.

Back-up blood samples will be collected for re-analysis in case of failure of the test measurement or for samples lost in transit. The samples will be appropriately stored and destroyed at study closure. Monitoring and auditing procedures defined/agreed by the External board (Sequre s.r.l. and Kilimo s.r l.) will be followed, in order to comply with GCP guidelines. This will include on-site checking of the case report forms (CRF) for completeness and clarity, cross-checking with source documents, and clarification of administrative matters.

Primary endpoints:

* To determine the safety, the maximum tolerated dose (MTD) and the RP2D of LNA-i-miR-221 using escalating doses in refractory multiple myeloma (MM) and advanced solid tumors for further investigations.
* To assess the safety and toxicity of LNA-i-miR-221

Secondary endpoints:

* PK analysis
* To preliminary explore the antitumor activity, the disease control, and the efficacy
* Biomodulatory activity A minimum/maximum number of 15/36 subjects will be enrolled in the study, according to expansion cohorts. All clinical data will be inserted on the Case Report Form (CRF) pages and all data can be extracted for the purpose of the ongoing analysis of the SRC and for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age ≥18 yrs
* Diagnosis of symptomatic multiple myeloma with measurable disease, i.e. detectable monoclonal component (MC) in the serum and/or urine.
* Patients with evidence of refractory disease according to IMWG criteria, who are either not suitable for bone marrow transplantation procedures or have relapsed after bone marrow transplantation and have failed at least three prior lines of therapy (10) (i.e. patients with lack of response or patients whose disease progresses on or within 60 days after the completion of last treatment).
* Histologically diagnosed stromal or epithelial solid tumors (clinically diagnosed HCC according to AASLD/EASLD guidelines).
* Patients with inoperable tumor(s) and no applicable curative therapy, not amenable to loco-regional therapy and/or codified standard systemic treatment, as established in the context of internationally accepted treatment guidelines for the various types of tumors that will be enrolled. One measurable target lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
* Life expectancy of at least three months according to physician evaluation
* ECOG 0-2
* Screening hematology, clinical chemistries, coagulation and urine analyses are not clinically significant and the following criteria are met:

  1. Platelets >75,000/mm3
  2. ANC >1000/mm3
  3. Hemoglobin > 8 g/dL
  4. Total and direct bilirubin < 2.5 mg/dl (except for clearly documented Gilbert's Syndrome)
  5. ALT and AST < 5 x ULN
  6. International normalized ratio (INR) <2.3 or prothrombin time (PT) <6 seconds above control
  7. Serum creatinine WNL and estimated by the Cockcroft-Gault formula or measured creatinine clearance rate > 40 ml/min
* Negative results on the following screening laboratory tests:

  1. urine or serum pregnancy test (for women of childbearing potential),
  2. human immunodeficiency virus (HIV) antibody.
* For men and women of childbearing potential, willingness to utilize adequate contraception and not become pregnant (or have their partner become pregnant) during the full course of the study.
* For female study participants, adequate birth control methods will be defined as: intrauterine device or double barrier contraception, i.e., condom plus diaphragm, condom or diaphragm plus spermicidal gel /foam
* For males study participants, adequate birth control methods will be defined as:

double barrier contraception, i.e., condom plus diaphragm; condom or diaphragm plus spermicidal gel/foam.

Note: Females who are not of childbearing potential must meet one of the following criteria:

1. Post-menopause - defined as one year without menses or follicle-stimulating hormone (FSH) of >40 U/mL
2. Surgical menopause - hysterectomy, bilateral oophorectomy, or bilateral tubal ligation
3. Pregnancy, breastfeeding

   * Subjects who participated to any other investigational drug trial within 30 days before enrollment to this trial
   * Severe liver dysfunction (Child-Pugh Class C or hepatic encephalopathy).
   * Serious medical or psychiatric illness, that may affect the correct participation to the trial
   * Concurrent social conditions (e.g. drug/alcohol abuse issue), that would potentially affect the correct participation to the trial New York Heart Association (NYHA) Class III or IV
   * cardiac disease, myocardial infarction within the past 6 months, unstable and/or symptomatic arrhythmia, or evidence of ischemia on ECG
   * Patients with active infections requiring systemic therapy are ineligible
   * Patients HIV positive or acquired immunodeficiency syndrome-related illness are ineligible
   * History of other malignancies within 3 years prior to study entry except for adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer or breast, low grade, early stage localized prostate cancer treated surgically with curative intent (TNM stage of T1a or T1b)
   * Voluntary written informed consent released before any study related procedure is performed. The consent may be withdrawn by the subject at any time without prejudice to future medical care.

Exclusion Criteria:

* Pregnancy,
* breastfeeding
* Subjects who participated to any other investigational drug trial within 30 days before enrollment to this trial
* Severe liver dysfunction (Child-Pugh Class C or hepatic encephalopathy).
* Serious medical or psychiatric illness, that may affect the correct participation to the trial
* Concurrent social conditions (e.g. drug/alcohol abuse issue), that would potentially affect the correct participation to the trial New York Heart Association (NYHA) Class III or IV
* cardiac disease, myocardial infarction within the past 6 months, unstable and/or symptomatic arrhythmia, or evidence of ischemia on ECG
* Patients with active infections requiring systemic therapy are ineligible
* Patients HIV positive or acquired immunodeficiency syndrome-related illness are ineligible
* History of other malignancies within 3 years prior to study entry except for adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer or breast, low grade, early stage localized prostate cancer treated surgically with curative intent (TNM stage of T1a or T1b)
* ECOG>2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2021-12-29 (Actual); Study Completion 2021-12-29 (Actual)

PRIMARY OUTCOMES:
Safety measured by adverse events To assess the toxicity of LNA-i-miR-221 | two years
  To assess the safety and toxicity of LNA-i-miR-221
The maximum tolerated dose (MTD) of LNA-i-miR-221 | two years
  The maximum tolerated dose (MTD) is the dose level below the dose level at which at least 2 out of 6 patients experience DLT.
The recommended phase II dose of LNA-i-miR-221 (RP2D) | two years
  recommended phase II dose of LNA-i-miR-221 (RP2D) using escalating doses for further evaluation

SECONDARY OUTCOMES:
To assess the Cmax of ascending doses of LNA-i-miR-221 | During first 6 days of dosing
  Peak Plasma Concentration of LNA-i-miR-221
To assess the Area under the plasma concentration versus time curve (AUC) of ascending doses of LNA-i-miR-221 | During first 6 days of dosing
  plasma concentration-time profile of LNA-i-miR-221
To assess the LNA-i-miR-221 clearance | During first 6 days of dosing
  the total body clearance of LNA-i-miR-221
To assess LNA-i-miR-221 biological half-life | During first 6 days of dosing
  t½, LNA-i-miR-221 apparent half-life
To assess the efficacy of LNA-i-miR-221 | Tumor response will be assessed after 30 (+/-1) days from the start of treatment
  Preliminary assessment of the clinical benefit and antitumoral activity of LNA-i-miR-221 based on RECIST V1.1 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Pierfrancesco Tassone, MD, Principal Investigator — Translational Medical Oncology Unit, AOU MaterDomini and Magna Graecia University
Locations (1):
- Center for Phase I Clinical Studies in Medical Oncology and Oncohematology - Translational Medical Oncology Unit, AOU MaterDomini and Magna Graecia University, Catanzaro, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Di Martino MT, Arbitrio M, Caracciolo D, Scionti F, Tagliaferri P, Tassone P. Dose-Finding Study and Pharmacokinetics Profile of the Novel 13-Mer Antisense miR-221 Inhibitor in Sprague-Dawley Rats. Mol Ther Nucleic Acids. 2020 Jun 5;20:73-85. doi: 10.1016/j.omtn.2020.01.036. Epub 2020 Feb 8. PMID 32146420
- [Background] Di Martino MT, Arbitrio M, Fonsi M, Erratico CA, Scionti F, Caracciolo D, Tagliaferri P, Tassone P. Allometric Scaling Approaches for Predicting Human Pharmacokinetic of a Locked Nucleic Acid Oligonucleotide Targeting Cancer-Associated miR-221. Cancers (Basel). 2019 Dec 19;12(1):27. doi: 10.3390/cancers12010027. PMID 31861748
- [Background] Gallo Cantafio ME, Nielsen BS, Mignogna C, Arbitrio M, Botta C, Frandsen NM, Rolfo C, Tagliaferri P, Tassone P, Di Martino MT. Pharmacokinetics and Pharmacodynamics of a 13-mer LNA-inhibitor-miR-221 in Mice and Non-human Primates. Mol Ther Nucleic Acids. 2016 Jun 21;5(6). doi: 10.1038/mtna.2016.36. PMID 27327137
- [Background] Franzoni S, Morbioli L, Turtoro A, Solazzo L, Greco A, Arbitrio M, Tagliaferri P, Tassone P, Di Martino MT, Breda M. Development and validation of bioanalytical methods for LNA-i-miR-221 quantification in human plasma and urine by LC-MS/MS. J Pharm Biomed Anal. 2020 Sep 5;188:113451. doi: 10.1016/j.jpba.2020.113451. Epub 2020 Jun 29. PMID 32659676
- [Background] Gulla A, Di Martino MT, Gallo Cantafio ME, Morelli E, Amodio N, Botta C, Pitari MR, Lio SG, Britti D, Stamato MA, Hideshima T, Munshi NC, Anderson KC, Tagliaferri P, Tassone P. A 13 mer LNA-i-miR-221 Inhibitor Restores Drug Sensitivity in Melphalan-Refractory Multiple Myeloma Cells. Clin Cancer Res. 2016 Mar 1;22(5):1222-33. doi: 10.1158/1078-0432.CCR-15-0489. Epub 2015 Nov 2. PMID 26527748
- [Background] Di Martino MT, Gulla A, Gallo Cantafio ME, Altomare E, Amodio N, Leone E, Morelli E, Lio SG, Caracciolo D, Rossi M, Frandsen NM, Tagliaferri P, Tassone P. In vitro and in vivo activity of a novel locked nucleic acid (LNA)-inhibitor-miR-221 against multiple myeloma cells. PLoS One. 2014 Feb 21;9(2):e89659. doi: 10.1371/journal.pone.0089659. eCollection 2014. PMID 24586944
- [Background] Franzoni S, Vezzelli A, Turtoro A, Solazzo L, Greco A, Tassone P, Di Martino MT, Breda M. Development and validation of a bioanalytical method for quantification of LNA-i-miR-221, a 13-mer oligonucleotide, in rat plasma using LC-MS/MS. J Pharm Biomed Anal. 2018 Feb 20;150:300-307. doi: 10.1016/j.jpba.2017.12.027. Epub 2017 Dec 15. PMID 29268195
- [Background] Di Martino MT, Gulla A, Cantafio ME, Lionetti M, Leone E, Amodio N, Guzzi PH, Foresta U, Conforti F, Cannataro M, Neri A, Giordano A, Tagliaferri P, Tassone P. In vitro and in vivo anti-tumor activity of miR-221/222 inhibitors in multiple myeloma. Oncotarget. 2013 Feb;4(2):242-55. doi: 10.18632/oncotarget.820. PMID 23479461
- [Background] Di Martino MT, Rossi M, Caracciolo D, Gulla A, Tagliaferri P, Tassone P. Mir-221/222 are promising targets for innovative anticancer therapy. Expert Opin Ther Targets. 2016 Sep;20(9):1099-108. doi: 10.1517/14728222.2016.1164693. Epub 2016 Mar 21. PMID 26959615
- [Background] Santolla MF, Lappano R, Cirillo F, Rigiracciolo DC, Sebastiani A, Abonante S, Tassone P, Tagliaferri P, Di Martino MT, Maggiolini M, Vivacqua A. miR-221 stimulates breast cancer cells and cancer-associated fibroblasts (CAFs) through selective interference with the A20/c-Rel/CTGF signaling. J Exp Clin Cancer Res. 2018 May 2;37(1):94. doi: 10.1186/s13046-018-0767-6. PMID 29716623
- [Background] Calura E, Bisognin A, Manzoni M, Todoerti K, Taiana E, Sales G, Morgan GJ, Tonon G, Amodio N, Tassone P, Neri A, Agnelli L, Romualdi C, Bortoluzzi S. Disentangling the microRNA regulatory milieu in multiple myeloma: integrative genomics analysis outlines mixed miRNA-TF circuits and pathway-derived networks modulated in t(4;14) patients. Oncotarget. 2016 Jan 19;7(3):2367-78. doi: 10.18632/oncotarget.6151. PMID 26496024
- [Derived] Tassone P, Di Martino MT, Arbitrio M, Fiorillo L, Staropoli N, Ciliberto D, Cordua A, Scionti F, Bertucci B, Salvino A, Lopreiato M, Thunarf F, Cuomo O, Zito MC, De Fina MR, Brescia A, Gualtieri S, Riillo C, Manti F, Caracciolo D, Barbieri V, Di Paola ED, Di Francesco AE, Tagliaferri P. Safety and activity of the first-in-class locked nucleic acid (LNA) miR-221 selective inhibitor in refractory advanced cancer patients: a first-in-human, phase 1, open-label, dose-escalation study. J Hematol Oncol. 2023 Jun 26;16(1):68. doi: 10.1186/s13045-023-01468-8. PMID 37365583
- See also: Volume 4 of "The rules governing medicinal products in the European Union" for human and veterinary use — https://ec.europa.eu/health/documents/eudralex/vol-4_en